CLINICAL TRIAL: NCT04087213
Title: Clinical Evaluation of the HemoCare™ Hemodialysis System for Home Nocturnal Hemodialysis
Brief Title: Study of HemoCare™ Hemodialysis System for Home Nocturnal Dialysis in Patients With ESRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deka Research and Development (Industry)
Collaborators: CVS Kidney Care LLC. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKPL-00057-001
Record Dates: First submitted 2019-08-30; First posted 2019-09-12 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-01

CONDITIONS: End-Stage Renal Disease
Keywords: HemoCare™ Hemodialysis System; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This is a prospective multi-center, open-label, single-arm, cross-over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- The HemoCare™ Hemodialysis System (Experimental): The HemoCare™ Hemodialysis System is intended for hemodialysis treatment, including short daily and nocturnal hemodialysis, of renal failure patients. The HemoCare™ Hemodialysis System is intended for use in chronic dialysis facilities, self-care dialysis facilities, or the home setting. All treatments must be prescribed by a physician and administered by a trained operator. Treatments must be performed under the supervision or assistance of a medical professional or a care partner who has been trained and deemed competent in the use of the device by the prescribing physician.
  Interventions: Device: HemoCare™ Hemodialysis System

INTERVENTIONS:
Device: HemoCare™ Hemodialysis System — The HemoCare™ Hemodialysis System is intended for hemodialysis treatment, including short daily and nocturnal hemodialysis, of renal failure patients. The HemoCare™ Hemodialysis System is intended for use in chronic dialysis facilities, self-care dialysis facilities, or the home setting. All treatments must be prescribed by a physician and administered by a trained operator. Treatments must be performed under the supervision or assistance of a medical professional or a care partner who has been trained and deemed competent in the use of the device by the prescribing physician.

SUMMARY:
This prospective multi-center, open-label, single-arm study intends to gather and evaluate safety data for the nocturnal use of the HemoCare™ Hemodialysis System.

DETAILED DESCRIPTION:
The HemoCare™ Hemodialysis System has been evaluated in previous clinical trials and is designed to perform hemodialysis (HD) in a clinic setting, in a self-care setting, or in a home environment for conventional HD, short daily HD or extended-duration HD therapy during the daytime or at night dependent on the users' lifestyle or work schedule. This multi-center, open-label, single-arm cross-over study is designed specifically to gather and evaluate safety data for the use of the HemoCare™ Hemodialysis System (including labeling and training tools) during home nocturnal (during sleeping hours based on the patient schedule) use. Nocturnal HD therapy was chosen as a treatment in this study because of the clinical and humanistic benefits associated with it. In addition, its risk profile, especially when performed in a home setting, may be greater than either existing conventional or short daily HD therapies. In this regard, establishing an acceptable safety profile for home nocturnal HD therapy should be sufficient evidence to support conventional and short daily HD home therapies with HemoCare™ Hemodialysis System.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with ESRD and are ≥ 18 years of age.
* Are in stable clinical condition as judged by the treating physician, and confirmed by medical history, physical exam, and laboratory testing for 30 days prior to enrollment.
* Have been receiving HD for at least 30 days prior to study enrollment, are expected to survive for at least 12 months and in the opinion of the Investigator are stable to start in the trial.
* Have been dialyzing in a supervised medical facility or at home for ≥ 3 times per week.
* Are willing to comply with the study requirements for training and therapy with HemoCare™ Hemodialysis System for the entire study treatment period.
* Understand English and can provide written informed consent (both the subject and care partner).
* Are judged by the Investigator to be suitable for Home HD (the Investigator deems that with appropriate training, the subject and/or care partner will be able to successfully cannulate and/or manage the vascular access during the Unassisted Home Evaluable Period).
* Have a stable functioning vascular access as judged by the treating physician.
* Have a weekly stdKt/Vurea ≥ 2.0, an equivalent URR ≥ 0.65, rated Kt/Vurea ≥ 1.0 on one occasion within 30 days prior to enrollment.

Exclusion Criteria:

* Are pre-scheduled for a living donor transplant within the next 6 months.
* Have a contraindication to heparin.
* Are currently participating in another interventional study.
* Have experienced an acute myocardial infarction with hospitalization, coronary artery bypass surgery, or acute coronary ischemia requiring angioplasty or stent insertion within 90 days of screening.
* Have ongoing NYHA Class III or IV heart failure.
* Have a significant psychiatric disorder or mental disability that could interfere with the subject's ability to provide informed consent and/or comply with study procedures.
* Have ongoing sepsis or bacteremia and currently require IV antibiotics.
* Have an allergy to polysulfone dialyzer.
* Current self-reported pregnancy, actively planning to become pregnant within the next 12 months, lactating, or not using medically acceptable means of contraception during the study.
* Subject with fluid overload due to intractable ascites secondary to liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dialysis Clinic, Inc - NJ, North Brunswick, New Jersey
  - The Rogosin Institute, New York, New York
  - Dialysis Clinic Inc. - Knoxville, Knoxville, Tennessee
  - Dialysis Clinic, Inc., Nashville, Tennessee
  - Wellbound South Austin, Austin, Texas
  - Wellbound North Austin, Austin, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Renal Data System. USRDS 2017 Annual Data Report: Atlas of End-Stage Renal Disease in the United States. Bethesda, MD: National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases; 2017
- [Background] Eloot S, Van Biesen W, Dhondt A, Van de Wynkele H, Glorieux G, Verdonck P, Vanholder R. Impact of hemodialysis duration on the removal of uremic retention solutes. Kidney Int. 2008 Mar;73(6):765-70. doi: 10.1038/sj.ki.5002750. Epub 2007 Dec 26. PMID 18160958
- [Background] Culleton BF, Walsh M, Klarenbach SW, Mortis G, Scott-Douglas N, Quinn RR, Tonelli M, Donnelly S, Friedrich MG, Kumar A, Mahallati H, Hemmelgarn BR, Manns BJ. Effect of frequent nocturnal hemodialysis vs conventional hemodialysis on left ventricular mass and quality of life: a randomized controlled trial. JAMA. 2007 Sep 19;298(11):1291-9. doi: 10.1001/jama.298.11.1291. PMID 17878421
- [Background] Rocco MV, Lockridge RS Jr, Beck GJ, Eggers PW, Gassman JJ, Greene T, Larive B, Chan CT, Chertow GM, Copland M, Hoy CD, Lindsay RM, Levin NW, Ornt DB, Pierratos A, Pipkin MF, Rajagopalan S, Stokes JB, Unruh ML, Star RA, Kliger AS; Frequent Hemodialysis Network (FHN) Trial Group; Kliger A, Eggers P, Briggs J, Hostetter T, Narva A, Star R, Augustine B, Mohr P, Beck G, Fu Z, Gassman J, Greene T, Daugirdas J, Hunsicker L, Larive B, Li M, Mackrell J, Wiggins K, Sherer S, Weiss B, Rajagopalan S, Sanz J, Dellagrottaglie S, Kariisa M, Tran T, West J, Unruh M, Keene R, Schlarb J, Chan C, McGrath-Chong M, Frome R, Higgins H, Ke S, Mandaci O, Owens C, Snell C, Eknoyan G, Appel L, Cheung A, Derse A, Kramer C, Geller N, Grimm R, Henderson L, Prichard S, Roecker E, Rocco M, Miller B, Riley J, Schuessler R, Lockridge R, Pipkin M, Peterson C, Hoy C, Fensterer A, Steigerwald D, Stokes J, Somers D, Hilkin A, Lilli K, Wallace W, Franzwa B, Waterman E, Chan C, McGrath-Chong M, Copland M, Levin A, Sioson L, Cabezon E, Kwan S, Roger D, Lindsay R, Suri R, Champagne J, Bullas R, Garg A, Mazzorato A, Spanner E, Rocco M, Burkart J, Moossavi S, Mauck V, Kaufman T, Pierratos A, Chan W, Regozo K, Kwok S. The effects of frequent nocturnal home hemodialysis: the Frequent Hemodialysis Network Nocturnal Trial. Kidney Int. 2011 Nov;80(10):1080-91. doi: 10.1038/ki.2011.213. Epub 2011 Jul 20. PMID 21775973
- [Background] Pauly RP, Gill JS, Rose CL, Asad RA, Chery A, Pierratos A, Chan CT. Survival among nocturnal home haemodialysis patients compared to kidney transplant recipients. Nephrol Dial Transplant. 2009 Sep;24(9):2915-9. doi: 10.1093/ndt/gfp295. Epub 2009 Jul 7. PMID 19584107
- [Background] Bernardo AA, Marbury TC, McFarlane PA, Pauly RP, Amdahl M, Demers J, Hutchcraft AM, Leypoldt JK, Minkus M, Muller M, Stallard R, Culleton BF. Clinical safety and performance of VIVIA: a novel home hemodialysis system. Nephrol Dial Transplant. 2017 Apr 1;32(4):685-692. doi: 10.1093/ndt/gfw044. PMID 27190336

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A required introduction to the HemoCare hemodialysis system and successful training for cannulation/ vascular access care at the study site for a minimum of 1-week prior to first home treatment (In-Facility Introduction Period).
Groups:
- Assisted Home Hemodialysis Then Unassisted Home Hemodialysis: Assisted: In-home treatment administered by a medical professional.
  Unassisted: In-home treatments either self-administered with the assistance of a care partner or administered by a care partner
Period: In-Facility Introduction
Arm/Group | Assisted Home Hemodialysis Then Unassisted Home Hemodialysis
Started | 36
Completed | 34
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Period: Transition Period A
Arm/Group | Assisted Home Hemodialysis Then Unassisted Home Hemodialysis
Started | 34
Completed | 34
Not Completed | 0
Period: Assisted Evaluable Period
Arm/Group | Assisted Home Hemodialysis Then Unassisted Home Hemodialysis
Started | 34
Completed | 29
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Personal reasons | 3
Period: Transition Period B
Arm/Group | Assisted Home Hemodialysis Then Unassisted Home Hemodialysis
Started | 29
Completed | 28
Not Completed | 1
Not completed — Renal Transplantation | 1
Period: Unassisted Home Evaluable Period
Arm/Group | Assisted Home Hemodialysis Then Unassisted Home Hemodialysis
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intent-To-Treat (ITT) Population: The ITT population was defined as all subjects who used HemoCare Hemodialysis System at least once during the Assisted Evaluable Period.
Arm/Group | Intent-To-Treat (ITT) Population
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 23
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: Adverse event (AE) rate per 100 HemoCare™ Hemodialysis System treatments during Assisted and Unassisted Home Evaluable Periods
Time Frame: 31 weeks
Population: The ITT population was defined as all subjects who used HemoCare Hemodialysis System at least once during the Assisted Evaluable Period.
Measure: Number; unit: Adverse Events per 100 Treatments
Groups:
- Assisted Evaluable Period: In-home treatment administered by a medical professional.
- Unassisted Home Evaluable Period: In-home HD treatments either self-administered with the assistance of a care partner or administered by a care partner
Arm/Group | Assisted Evaluable Period | Unassisted Home Evaluable Period
Number analyzed (Participants) | 34 | 28
Adverse Events per 100 Treatments | 16.1 | 11.6

2. Primary Outcome: Primary Performance Endpoint
Description: Weekly stdKt/Urea was calculated from pre- and post-dialysis urea levels during each evaluable period. Blood samples were obtained every two weeks during each Evaluable Period. For the primary performance endpoint, 'success' is defined as a subject who has all stdKt/Vurea measures in an evaluable period greater than or equal to 2.0.
Time Frame: 31 weeks
Population: Weekly stdKt/Vurea collected from the Intent-To-Treat (ITT) Population
Measure: Number (90% Confidence Interval); unit: Percentage of subjects with Kt/V ≥ 2.0
Arm/Group | Assisted Evaluable Period | Unassisted Home Evaluable Period
Number analyzed (Participants) | 34 | 28
Percentage of subjects with Kt/V ≥ 2.0 | 1 [0.92 to 1.00] | 1 [0.90 to 1.00]

3. Secondary Outcome: The Total Number of AEs and SAEs (Anticipated, Unanticipated, and Device Related)
Description: Number of anticipated and unanticipated AEs and SAEs during each Evaluable Period including number of device-related AEs and SAEs.
Time Frame: 31 weeks
Population: Adverse Events reported by the Intent-To-Treat (ITT) Population
Measure: Number; unit: events
Arm/Group | Assisted Evaluable Period | Unassisted Home Evaluable Period
Number analyzed (Participants) | 34 | 28
events
  Total Adverse Events | 204 | 139
  Anticipated Non-Serious AE | 148 | 11
  Anticipated Serious AE | 5 | 2
  Unanticipated Non-Serious AE | 49 | 26
  Unanticipated Serious AE | 2 | 0
  Device-Related Non-Serious AE | 27 | 7
  Device-Related Serious AE | 0 | 0
  Unanticipated Device-Related Non-Serious AE | 0 | 0
  Unanticipated Device-Related Serious AE | 0 | 0

4. Secondary Outcome: The Number of Decreased and Increased Post-dialysis Serum Phosphorus Levels
Description: The number of decreased serum phosphorus defined as at least 1 post-dialysis serum phosphorus level < 2.2 mg/dL , the number of elevated serum phosphorous defined as a least 1 post-dialysis serum phosphorus level > 5.5 mg/dL, will each be compared between Evaluable Periods with exact McNemar's tests.
Time Frame: 31 weeks
Population: Intent-To-Treat (ITT) Population
Measure: Number; unit: occurrence of event
Arm/Group | Assisted Evaluable Period | Unassisted Home Evaluable Period
Number analyzed (Participants) | 34 | 28
occurrence of event
  Decreased serum phosphorous | 48 | 32
  Increased serum phosphorous | 0 | 2

5. Secondary Outcome: The Number of Decreased and Increased Post-dialysis Serum Potassium During Each Evaluable Period.
Description: The number of decreased serum potassium defined as at least 1 post-dialysis serum potassium level of < 3.5 meq/L , and the number of elevated serum potassium defined as at least 1 post-dialysis serum potassium level of > 5.9 meq/L, will each be compared between Evaluable Periods with exact McNemar's tests.
Time Frame: 31 weeks
Population: Intent-To-Treat (ITT) Population
Measure: Number; unit: events
Arm/Group | Assisted Evaluable Period | Unassisted Home Evaluable Period
Number analyzed (Participants) | 34 | 28
events
  Decreased serum potassium | 43 | 24
  Elevated serum potassium | 0 | 1

6. Secondary Outcome: Weight Change and Fluid Removed Comparison Between Evaluable Periods
Description: HemoCare Ultrafiltration Comparison by Evaluable Period was determined by the following:
  Discrepancy between Weight Change and Net UF removed = Weight change - Net UF Removed
  Weight change = Ending weight - Starting weight (measured by digital weight scale).
  Net Ultrafiltration Removed = total UF removed - prime & rinseback, reported by the HemoCare system.
  Note: One kilogram (kg) = one liter (L) of fluid
Time Frame: 31 weeks
Population: Intent-To-Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Assisted Evaluable Period | Unassisted Home Evaluable Period
Number analyzed (Participants) | 34 | 28
L | 0.1 (3.5) | 0.1 (1.1)

ADVERSE EVENTS:
Time Frame: During the study period - from the time of enrollment until the end of participation in the study (31 weeks).
Description: All Adverse Events and Serious Adverse Events were recorded, regardless of relatedness.
Arm/Group | Assisted Evaluable Period | Unassisted Home Evaluable Period
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/34 | 2/28
Other Adverse Events (participants affected / at risk) | 31/34 | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assisted Evaluable Period (N=34) | Unassisted Home Evaluable Period (N=28)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypervolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assisted Evaluable Period (N=34) | Unassisted Home Evaluable Period (N=28)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Edema (General disorders) | 2 (3) | 0 (0)
Edema peripheral (General disorders) | 3 (3) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 (7) | 2 (6)
Arteriovenous fistula site hematoma (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Vascular access site hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 0 (0)
Blood calcium decreased (Investigations) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)
Blood phosphorus decreased (Investigations) | 2 (2) | 3 (3)
Blood phosphorus increased (Investigations) | 0 (0) | 2 (3)
Blood potassium increased (Investigations) | 2 (2) | 0 (0)
Hemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 4 (5) | 4 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (9) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (13) | 6 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 7 (8) | 4 (7)
Headache (Nervous system disorders) | 8 (10) | 6 (15)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Thrombosis in device (Product Issues) | 2 (2) | 2 (3)
Hemorrhage (Vascular disorders) | 8 (25) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT04087213/Prot_SAP_000.pdf